CLINICAL TRIAL: NCT03024268
Title: MitraClip® and Hemodynamic Effects of Relevant Iatrogenic Atrial Septum Defect Closure - Evaluation of Morphologic and Functional Changes in a Randomized Setting
Brief Title: MitraClip® and Hemodynamic Effects of Relevant Iatrogenic Atrial Septum Defect Closure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Heart Center Leipzig - University Hospital (Other)
Responsible Party: Principal Investigator, Philipp Lurz, Clinical Investigator, Professor, Managing Senior Physician, Heart Center Leipzig - University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MITHRAS
Record Dates: First submitted 2016-12-29; First posted 2017-01-18 (Estimated); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: Mitral Valve Insufficiency; Heart Septal Defects, Atrial
MeSH Terms: conditions — Mitral Valve Insufficiency; Heart Septal Defects, Atrial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A: interventional closure of iASD (Experimental): Interventional closure of iASD (n=40) with an Figulla Flex Occluder (Occlutech)
  Interventions: Device: Figulla Flex Occluder (Occlutech)
- B: no intervention (No Intervention): Best medical supportive care (n=40)

INTERVENTIONS:
Device: Figulla Flex Occluder (Occlutech) — Interventional closure of the iASD with an Figulla Flex Occluder (Occlutech)
  Arms: A: interventional closure of iASD

SUMMARY:
Aim of this prospective trial is to assess the hemodynamic effects of a MitraClip procedure caused iatrogenic arterial septal defect (iASD) and the functional changes after interventional iASD closure in a randomized setting.

DETAILED DESCRIPTION:
Transcatheter mitral valve repair with the MitraClip system is a therapeutic alternative to surgery in selected high-risk patients. Clip placement requires interatrial transseptal puncture and meticulous manipulation of the steerable sheath. There is evidence that the persistence of a relevant iASD after MitraClip is associated with worse clinical outcomes and increased mortality.

The purpose of this study is to investigate, if the interventional closure of an persistant hemodynamic relevant iASD 30 days after MitraClip implantation, has favorable effects on clinical outcome. Eligible patients, after obtaining written informed consent, are 1:1 randomized either in group A (interventional occlusion of iASD) or group B (best supportive care).

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Previous MitraClip implantation
* Persistent relevant iASD 30 days after MitraClip intervention

Exclusion Criteria:

* Unsuccessful MitraClip implantation
* No relevant iASD 30 days after MitraClip intervention
* Unstable angina in the previous 4 weeks
* Valvular heart disease (aortic, tricuspid or pulmonary valve) planed for surgery or interventional therapy
* Constrictive pericarditis / restrictive cardiomyopathies
* Pericardial effusion planed for surgery or interventional therapy
* Coagulation disorders
* Malignant disease with a life expectance < 12 months
* Pregnancy
* Participation in another study
* iASD diameter > 38 mm
* Aortic minimum distance of the iASD < 5 mm
* Thrombus in left atrial appendage
* Venous access impossible with a 24 French catheter system
* Presence of an inferior vena cava filter

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2020-09 (Actual); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Change in Exercise tolerance: 6 minute walking test | baseline, 3 and 6 months

SECONDARY OUTCOMES:
Change in New York Heart Association Functional Classification assessment | baseline, 3 and 6 months
  Changes in New York Heart Association Functional Classification
Changes in Echocardiography: bi ventricular function (2D and 3D) | baseline, 3 and 6 months
Changes in Echocardiography: assessment of left atrium (2D and 3D) | baseline, 3 and 6 months
Changes in Echocardiography: assessment of heart valves | baseline, 3 and 6 months
Changes in Echocardiography: strain using speckle tracking | baseline, 3 and 6 months
Changes in Echocardiography: evaluation of iatrogenic ASD (2D and 3D) | baseline, 3 and 6 months
Heart insufficiency bio markers | baseline and 6 months
Changes in Cardiac MRI: bi ventricular function | baseline and 6 months
Changes in Cardiac MRI: left ventricular longitudinal strain | baseline and 6 months
Changes in Cardiac MRI: left ventricular circumferential strain | baseline and 6 months
Changes in Cardiac MRI: flow measurements in main pulmonary artery and aorta | baseline and 6 months
Evaluation of hospitalisation rate | baseline, 3, 6 and 12 months
  Telephone
Evaluation of mortality | baseline, 3, 6 and 12 months
  Telephone
Combined endpoint (hospitalisation and mortality) | baseline, 3, 6 and 12 months
  Telephone; Combined Endpoint of hospitalisation and mortality. For analysis the first event is counted regardless of severity.
Changes in quality of life in "Minnesota Living with Heart Failure" questionnaire | baseline and 6 months
Changes in quality of life in "Short Form - 36" questionnaire | baseline and 6 months

OTHER OUTCOMES:
Acute changes in right and left ventricular pressures during interventionell ASD closure | immediately before and immediately after ASD closure

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Lurz, MD, PhD, Principal Investigator — Heart Center of the University Leipzig; Stephan Blazek, MD, Study Chair — Heart Center of the University Leipzig
Locations (1):
- Heart Center of the University Leipzig, Leipzig, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Blazek S, Unterhuber M, Rommel KP, Kresoja KP, Kister T, Besler C, Fengler K, Rosch S, Daehnert I, Thiele H, Lurz P, von Roeder M. Fate of iatrogenic atrial septal defects following mitral transcatheter edge-to-edge repair - a subanalysis of the MITHRAS trial. Int J Cardiovasc Imaging. 2023 Mar;39(3):519-530. doi: 10.1007/s10554-022-02750-5. Epub 2022 Nov 13. PMID 36371488
- [Derived] Lurz P, Unterhuber M, Rommel KP, Kresoja KP, Kister T, Besler C, Fengler K, Sandri M, Daehnert I, Thiele H, Blazek S, von Roeder M. Iatrogenic Atrial Septal Defects Following Transcatheter Mitral Valve Repair and Implications of Interventional Closure. JACC Cardiovasc Interv. 2021 Dec 27;14(24):2685-2694. doi: 10.1016/j.jcin.2021.09.023. PMID 34949392